CLINICAL TRIAL: NCT04716556
Title: TranSfUsion of coNvalescent plAsma for the Early Treatment of pneuMonIa Due to SARS-CoV2 (TSUNAMI Study): a Multicenter Open Label Randomized Control Trial
Brief Title: TranSfUsion of coNvalescent plAsma for the Early Treatment of pneuMonIa in COVID-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Superiore di Sanità (Other)
Collaborators: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other); Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Principal Investigator, Elena Toschi, Research Coordinator, Istituto Superiore di Sanità
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSUNAMI
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Covid19; Coronavirus Infection; Pneumonia, Viral
Keywords: plasma
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Pneumonia, Viral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Therapy+Convalescent Plasma (Experimental): Patients will receive standard therapy + 200-300 ml of convalescent plasma for a maximum of 3 times in 5 days, according to clinical conditions.
  Interventions: Biological: Convalescent plasma
- Standard Therapy (No Intervention): Patients will receive standard therapy for the treatment of SARS-CoV2 infection, according to AIFA indications

INTERVENTIONS:
Biological: Convalescent plasma — Convalescent plasma will be collected by healthy donors, recovered by COVID19 and, after standard preparation and dosage of neutralizing antibodies, it will be administered to patients with SARS-CoV2 pneumonia
  Arms: Standard Therapy+Convalescent Plasma

SUMMARY:
This is a multicenter open-label randomized study for the early treatment of pneumonia due to SARS-COV2 with transfusion of convalescent plasma.

Patients with pneumonia due to SARS-CoV-2 will be randomized to receive or not convalescent plasma collected by recovered patients with previous diagnosis of COVID19

DETAILED DESCRIPTION:
This is a multicenter open-label randomized study for the early treatment of pneumonia due to SARS-COV2 with transfusion of convalescent plasma.

Patients with SARS-CoV2 pneumonia not requiring mechanical ventilation (both non invasive and invasive) will be randomized to receive or not convalescent plasma.

Patients in the plasma group will receive 200-300 ml of plasma collected by recovered patients with previous diagnosis of COVID19, plus standard therapy; Patients in the control group will receive the standard therapy. A rescue therapy will be allowed in case of clinical worsening.

Patients will be followed until day n30 from randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* adult patients with positive RT-PCR test for SARS-CoV2 (nasal swabs or lower respiratory tract sample), diagnosed with pneumonia (<= 10 days) according to the following definitions:

  * Suggestive radiological imaging (CT, RX, ultrasound);
  * Respiratory failure not fully explained by heart failure or fluid overload;
  * PaO2/FiO2 200-350 mmHg;
  * Signed informed consent

Exclusion Criteria:

* need of non invasive or invasive mechanical ventilation at the time of randomization;
* PaO2/FiO2 <200;
* patients with hypersensitivity or allergic reaction to blood products or immunoglobulins;
* patients who expressly refuse to adhere the clinical study;
* use of IL-6 Receptor inhibitors, IL-1 inhibitors, JAK inhibitors, TNF inhibitors;
* patients participating to other clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Number of patients who meet invasive mechanical ventilation or death | at 30 days
  Number of patients who meet invasive mechanical ventilation defined as PaO2/FiO2 <150 or death

SECONDARY OUTCOMES:
Mortality rates | 30 days
  Mortality rates at 30 days
Time to invasive mechanical ventilation or death | 30 days
  Days from randomization to invasive mechanical ventilation or death
Time to virologic recover | 30 days
  Days from randomization to virologic recover (defined as 2 consecutive negative nasopharynx tests)
Hospitalization time | 30 days
Adverse events | 30 days
  occurrence of Adverse events

OTHER OUTCOMES:
Evaluation of CD4/CD8 ratio | 14 days

CONTACTS AND LOCATIONS:
Locations (48):
- Italy (48):
  - SOD Clinica Malattie Infettive Tropicali, Parassitologia, Epatiti Croniche - AOU Ospedali Riuniti di Ancona, Ancona
  - Ospedale di Arezzo, Arezzo
  - Clinica Malattie Infettive, Università degli Studi di Bari, Bari
  - Ospedale Papa Giovanni XXIII-Dip. emergenza, Urgenza e area critica, Bergamo
  - UOC Malattie Infettive - AOU Bologna, Bologna
  - UO PID Tossicologia Applicata - Dip. Scienze Biomediche e Biotecnologiche - Università di Catania - AOU Policlinico Vittorio Emanuele, Catania
  - Ospedale Città di Castello, Città di Castello
  - Ospedale di Empoli, Empoli
  - UOC Malattie Infettive - ASUR Marche Area Vasta 4, Fermo
  - UOC Malattie Infettive - AOU Ferrara, Ferrara
  - Ospedale Santa Maria Annunziata, Florence
  - SOD Malattie Infettive e Tropicali - AOU Careggi, Florence
  - Dip.Medicina Clinica e Sperimentale - Policlinico "Riuniti" di Foggia, Foggia
  - Nuovo Ospedale S. Giovanni Battista Usl Umbria2, Foligno
  - U.O.C. Malattie Infettive ASL Frosinone, Frosinone
  - U.O. Malattie Infettive IRCCS-Ospedale Policlinico San Martino, Genova
  - Ospedale di Grosseto, Grosseto
  - ASL 5 Spezzina - SC Malattie Infettive, La Spezia
  - ASST Lecco - Malattie Infettive, Lecco
  - Ospedale di Livorno, Livorno
  - Ospedale di Lucca, Lucca
  - S.C. Pneumologia e Utir ASST Mantova - Ospedale Carlo Poma, Mantova
  - Ospedale Dell'Angelo - UOC Malattie Infettive, Mestre
  - ASST Santi Paolo e Carlo, Milan
  - Ospedale Luigi Sacco, Milan
  - SC Malattie Infettive ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Ospedale San Gerardo, Monza
  - Malattie Infettive - AOU Federico II di Napoli, Napoli
  - UOC Malattie Infettive ad indirizzo Respiratorio - PO Cotugno - AORN "Dei Colli", Napoli
  - UOC Malattie Infettive e Tropicali - AOU Policlinico, Palermo
  - Dip. Medicina Diagnost. e Servizi Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliero-Universitaria di Perugia, Perugia
  - UOC Malattie Infettive - Azienda Ospedali Riuniti Marche Nord, Pesaro
  - AOU Pisana, Pisa
  - Ospedale Pistoia, Pistoia
  - Ospedale Prato, Prato
  - Malattie Infettive Ravenna, Ravenna
  - UOC Malattie Infettive - AUSL Reggio Emilia, Reggio Emilia
  - Malattie Infettive - Rimini Forlì Cesena, Rimini
  - Campus Bio Medico - UO Anestesia e Rianimazione, Roma
  - ASL 1 Imperiese - SC Malattie Infettive, Sanremo
  - ASL 2 Savonese - SC Malattie Infettive, Savona
  - Ospedale di Siena, Siena
  - Ospedale di Sondrio - dipartimento di Medicina, Sondrio
  - AOU di Terni, Terni
  - Ospedale Ca Foncello - UOC Malattie Infettive, Treviso
  - A.O. Integrata Università di Verona, Verona
  - Ospedale Viareggio, Viareggio

REFERENCES:
- [Derived] Menichetti F, Popoli P, Puopolo M, Spila Alegiani S, Tiseo G, Bartoloni A, De Socio GV, Luchi S, Blanc P, Puoti M, Toschi E, Massari M, Palmisano L, Marano G, Chiamenti M, Martinelli L, Franchi S, Pallotto C, Suardi LR, Luciani Pasqua B, Merli M, Fabiani P, Bertolucci L, Borchi B, Modica S, Moneta S, Marchetti G, d'Arminio Monforte A, Stoppini L, Ferracchiato N, Piconi S, Fabbri C, Beccastrini E, Saccardi R, Giacometti A, Esperti S, Pierotti P, Bernini L, Bianco C, Benedetti S, Lanzi A, Bonfanti P, Massari M, Sani S, Saracino A, Castagna A, Trabace L, Lanza M, Focosi D, Mazzoni A, Pistello M, Falcone M; TSUNAMI Study group. Effect of High-Titer Convalescent Plasma on Progression to Severe Respiratory Failure or Death in Hospitalized Patients With COVID-19 Pneumonia: A Randomized Clinical Trial. JAMA Netw Open. 2021 Nov 1;4(11):e2136246. doi: 10.1001/jamanetworkopen.2021.36246. PMID 34842924